CLINICAL TRIAL: NCT04576897
Title: Non-invasive Evaluation of Portal Hypertension in Patients With Compensated Advanced Chronic Liver Disease by Liver Stiffness Measurement Using Liver Incytes
Brief Title: Velacur by Sonic Incytes for Portal Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Sonic Incytes (Industry)
Responsible Party: Principal Investigator, Samer Gawrieh, Professor of Clinical Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LI for Portal Hypertenstion; 2009698702 (Other: Indiana University IRB)
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Results first posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Portal Hypertension; Chronic Advanced Liver Disease
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Intervention Model Description: All participants will undergo quantitative ultrasound with Velacur by Sonic Incytes by a certified technician.
Masking Description: This is an open label study in that all participants will receive the same study procedures. Participants only receive this Velacur intervention if they are enrolled in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Velacur by Sonic Incytes (Experimental): Patients with compensated advanced chronic liver disease (cACLD) who have not undergone liver transplantation will be scanned with Velacur.
  Interventions: Diagnostic Test: Velacur

INTERVENTIONS:
Diagnostic Test: Velacur — Ultrasound elasticity imaging

SUMMARY:
This is a cross sectional study that evaluates the relationship between LSM (liver stiffness measurement) by Liver Incytes in patients with cACLD (compensated advanced chronic liver disease) and manifestations of portal hypertension.

DETAILED DESCRIPTION:
The purpose of this study is to assess the severity of portal hypertension in people with compensated advanced chronic liver disease (cACLD) who have not undergone liver transplant by measuring liver stiffness with the Liver Incytes device (Velacur) and comparing the performance of LSM (liver stiffness measurement) via Velcaur and transient elastography via FibroScan to esophageal varices.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older
2. Ability to provide informed consent
3. Planned standard of care upper endoscopy to screen for varices
4. Planned standard of care transjugular liver biopsy with portal pressure measurement

Exclusion Criteria:

1. Inability or refusal to provide informed consent
2. Fasting for less than three hours prior to the scan
3. Subject is a pregnant or lactating female
4. Subject with current, significant alcohol consumption
5. Patients with a pacemaker or defibrillator
6. Acute hepatitis defined as AST/ALT > 500 U/L
7. Ascites
8. post liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samer Gawrieh, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Division of Gastroenterolgy and Hepatology, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 participants enrolled in the study. The images from the Velacur device for all of the subjects were reviewed by the company. Only 33 of the enrolled participants had a valid Velacur study so results are reported only for these 33 participants. The remaining 37 participants were considered to have withdrawn from the study.
Pre-assignment Details: 70 participants enrolled in the study. The images from the Velacur device for all of the subjects were reviewed by the company. Only 33 of the enrolled participants had a valid Velacur study so results are reported only for these 33 participants. The remaining 37 participants were considered to have withdrawn from the study.
Groups:
- Liver Incytes: Patients with compensated advanced chronic liver disease (cACLD) who have not undergone liver transplantation will be scanned with Liver Incytes.
  Liver Incytes: Ultrasound elasticity imaging
Period: Overall Study
Arm/Group | Liver Incytes
Started | 70
Completed | 33
Not Completed | 37
Not completed — 37 scans were determined by the sponsor to be invalid. | 37

BASELINE CHARACTERISTICS:
Population: A total of 33 people underwent both Velacur and transient elastography via FibroScan and had results considered to be reliable
Groups:
- Liver Incytes: Patients with compensated advanced chronic liver disease (cACLD) who have not undergone liver transplantation will be scanned with Liver Incytes.
Arm/Group | Liver Incytes
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33
Velacur, liver stiffness [Mean (Standard Deviation); unit: kPa] | 9.9 (3.4)
Velacur, liver steatosis [Mean (Standard Deviation); unit: dB/m] | 313 (76)
transient elastography via FibroScan, liver stiffness [Mean (Standard Deviation); unit: kPa] | 37.8 (24.1)
transient elastography via FibroScan, liver steatosis [Mean (Standard Deviation); unit: dB/m] | 262 (73)

OUTCOME MEASURES:

1. Primary Outcome: Liver Stiffness Measurements for Participants With Compensated Advanced Chronic Liver Disease With and Without Esophageal Varices Upon Esophagogastroduodenoscopy (EGD)
Description: Comparing the performance of Velacur by Sonic Incytes to transient elastography via FibroScan® in the same patient population to determine if either test is more accurate in correlating with compensated advanced chronic liver disease (cACLD) for participants with and without esophageal varices.
Time Frame: one day
Measure: Mean (Standard Deviation); unit: kPa
Groups:
- Participants Without Evidences of Esophageal Varices; Participants With Evidence of Esophageal Varices: Patients with compensated advanced chronic liver disease (cACLD) who have not undergone liver transplantation will be scanned with Velacur by Sonic Incyes and transient elastography via FibroScan. All participants will have also undergone esophagogastroduodenoscopy (EGD).
  Results will be compared for participants with and without varices found in the EGD.
Arm/Group | Participants Without Evidences of Esophageal Varices | Participants With Evidence of Esophageal Varices
Number analyzed (Participants) | 10 | 23
kPa
  liver stiffness with Velacur | 9.6 (3.9) | 10.1 (3.2)
  liver stiffness with FibroScan | 26.5 (21.9) | 43.3 (23.5)

2. Primary Outcome: Platelet Count for Participants With Compensated Advanced Chronic Liver Disease
Description: Comparing the platelet count in the same patient population to determine Velacur's accuracy in correlating with compensated advanced chronic liver disease (cACLD) for participants with and without esophageal varices
Time Frame: one day
Measure: Mean (Standard Deviation); unit: in 100000 per microliter of blood
Groups:
- Participants With Evidence of Esophageal Varices: Patients with compensated advanced chronic liver disease (cACLD) who have not undergone liver transplantation will be scanned with Velacur. These participants have undergone esophagogastroduodenoscopy (EGD) with evidence of esophageal varices.
- Participants Without Evidence of Esophageal Varices: Patients with compensated advanced chronic liver disease (cACLD) who have not undergone liver transplantation will be scanned with Velacur. These participants have undergone esophagogastroduodenoscopy (EGD) without evidence of esophageal varices.
Arm/Group | Participants With Evidence of Esophageal Varices | Participants Without Evidence of Esophageal Varices
Number analyzed (Participants) | 23 | 10
in 100000 per microliter of blood | 91.2 (37.7) | 138 (71)

3. Other Pre Specified Outcome: Correlation of Velacur Measurements to Non-Invasive Blood Markers for Predicting Advanced Fibrosis
Description: This was initially included in our study protocol as an outcome measurement. However, we realized that these markers were not being routinely collected and the data are simply not available. Therefore, no outcome data are or can be included for this measurement.
Time Frame: one day
Population: During the course of this study, we realized that these markers were not being routinely collected and the data are simply not available. Therefore, no outcome data are or can be included for this measurement
Arm/Group | Participants Without Evidences of Esophageal Varices | Participants With Evidence of Esophageal Varices
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of study participation. This is a minimal risk study with only one study visit lasting less than one hour.
Description: The definition of adverse event utilized in this trial correlates with the clincialtrials.gov definition of adverse events.
Groups:
- Liver Incytes: Patients with compensated advanced chronic liver disease (cACLD) who have not undergone liver transplantation will be scanned with Liver Incytes.
  No adverse events were reported in this minimal risk study.
Arm/Group | Liver Incytes
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT04576897/Prot_004.pdf
  • Statistical Analysis Plan (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT04576897/SAP_005.pdf